CLINICAL TRIAL: NCT06913582
Title: Chang Gung Medical Foundation Institutional Review Board
Brief Title: The Effectiveness of Distance Yoga Learning in Improving Ma-ternal Pandemic-related Depression and Stress During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wen-Ping Lee, Head Nurse, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Kate65.0220
Record Dates: First submitted 2025-03-12; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Pregnancy Related
Keywords: distance yoga; pandemic; depression and stress; pregnancy
MeSH Terms: conditions — Depression | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: quasi-experimental design with experimental and control group.
Masking Description: First-time mothers between 20 and 26 weeks of pregnancy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experiment (Experimental): A 12-week pregnancy yoga program was delivered to experimental group (n=30) including one weekly 60-minute remote online yoga class and followed by 2 times of DVD yoga exercise.
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Behavioral: Yoga — A 12-week pregnancy yoga program was delivered to experimental group (n=30) including one weekly 60-minute remote online yoga class and followed by 2 times of DVD yoga exercise.

SUMMARY:
The goal of this quasi-experimental study design is to explore the effects of distance yoga learning in improving depression and pregnancy stress in pregnant women during the pandemic disease. The main questions which aim to answer are:

1. hypothesis1 - Distance yoga learning can decrease depression during pregnancy.
2. hypothesis2 -Distance yoga learning can decrease pregnancy stress. The experimental group received a 12-week pregnancy yoga program, including one weekly 60-minute distance yoga class and followed by 2 times of DVD yoga exercise at home while the control group received only routine nursing care.

DETAILED DESCRIPTION:
This is a quasi-experimental study design for primiparous women in the obstetrics and gynecology department of a regional hospital as the research subjects. This study received ethical approval from the hospital and all participants provided written informed consent. After the researcher took convenience samples and explained the research purpose in the prenatal parent classroom, they were assigned to the experimental group and the control group according to the wishes of the cases. Pregnant women in the experimental group received routine prenatal care guidance and yoga exercises three times a week, while the control group only received routine pre-natal guidance and the differences between the two groups were compared.

The sample size was estimated using G-power 3.1.9.2 software. The sample size was estimated to be 52 participants. Assuming the attrition rate was 20%, there were 32 people in the experimental group and the control group making a total of 64 participants.

During the study, one participant in the experimental group had premature delivery due to early water rupture, and the other one was hospitalized for tocolysis due to frequent uterine contractions and therefore withdrew from the experiment, resulting in a loss of 2 samples. For control group, one participant was admitted to the hospital for tocolysis due to prepartum hemorrhage and was withdrew from the study. Therefore, a total of 61 participants completed the study .

ELIGIBILITY:
Inclusion Criteria:

* First-time mothers between 20 and 26 weeks of pregnancy.
* normal fetus with a singleton.
* no history of smoking, drinking, or drug abuse.
* no bleeding during pregnancy.
* no related high-risk complications during pregnancy (such as high blood pressure, preeclampsia, gestational diabetes, heart dis-ease, etc.).
* no early abortion symptoms.
* Able to move normally.
* Able to listen, speak, read and write Chinese.
* Able to participate in the research and cooperate in completing the questionnaire.

Exclusion Criteria:Exclusion conditions (any one)

* Multiparous women.
* First-time mothers with pregnancy >26 weeks.
* Multiple births.
* Symptoms of bleeding or early miscarriage.
* Related high-risk pregnancy complications.

Ages: 22 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
demographic data and exercise history of two groups | 12 months
  Basic characteristics: Basic personal information included age, height, religious beliefs, marital status, education, daily activities, past medical history, etc. Obstetric variable information included weeks of pregnancy, pre-pregnancy weight, weight gained during pregnancy, and exercise before and during pregnancy, etc.
The change of depression status of two groups | 12 months
  Edinburgh Postnatal Depression Scale(EPDS): The Edinburgh Postnatal Depression Scale is used to measure prenatal and postpartum depressed mood. There are 10 questions in total, each question is scored on a 4-point scale. According to the order of each option, the first, second and fourth items are scored from 0 to 3 points, the other items are scored from 3 to 0 points, and the total score is from 0 to 30 points. The levels of scale were as follows: 0-9 points: low risk, usually no further psychological intervention is needed; 10-12 points: medium risk, further evaluation and observation are recom-mended; 13 points and above: high risk, comprehensive psychological evaluation and possible intervention measures should be carried out. The higher the score of pregnant women, the more severe the prenatal depression is.
Stress during pregnancy of two groups | 12 months
  Pregnancy Stress Rating Scale (PSRS): The "Pregnancy Stress Scale" developed by Chen, Huang, and Ka in 1991 and revised it into a new version of the "Pregnancy Stress Scale" by Chen was used in this study. The scale has five factors; it mainly measures the psychological stress experienced by women during pregnancy. There are 36 questions in total with the Likert five-point scoring method totaling score of 180 points. The higher the score, the greater the stress during pregnancy. The new version of the "Pregnancy Stress Scale" has good internal consistency (α=.92) and 2-week test-retest reliability (α=.82).

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nazzari S, Pili MP, Gunay Y, Provenzi L. Pandemic babies: A systematic review of the association between maternal pandemic-related stress during pregnancy and infant development. Neurosci Biobehav Rev. 2024 Jul;162:105723. doi: 10.1016/j.neubiorev.2024.105723. Epub 2024 May 16. PMID 38762129
- [Result] Lokken EM, Huebner EM, Taylor GG, Hendrickson S, Vanderhoeven J, Kachikis A, Coler B, Walker CL, Sheng JS, Al-Haddad BJS, McCartney SA, Kretzer NM, Resnick R, Barnhart N, Schulte V, Bergam B, Ma KK, Albright C, Larios V, Kelley L, Larios V, Emhoff S, Rah J, Retzlaff K, Thomas C, Paek BW, Hsu RJ, Erickson A, Chang A, Mitchell T, Hwang JK, Erickson S, Delaney S, Archabald K, Kline CR, LaCourse SM, Adams Waldorf KM; Washington State COVID-19 in Pregnancy Collaborative. Disease severity, pregnancy outcomes, and maternal deaths among pregnant patients with severe acute respiratory syndrome coronavirus 2 infection in Washington State. Am J Obstet Gynecol. 2021 Jul;225(1):77.e1-77.e14. doi: 10.1016/j.ajog.2020.12.1221. Epub 2021 Jan 27. PMID 33515516
- [Result] Zambrano LD, Ellington S, Strid P, Galang RR, Oduyebo T, Tong VT, Woodworth KR, Nahabedian JF 3rd, Azziz-Baumgartner E, Gilboa SM, Meaney-Delman D; CDC COVID-19 Response Pregnancy and Infant Linked Outcomes Team. Update: Characteristics of Symptomatic Women of Reproductive Age with Laboratory-Confirmed SARS-CoV-2 Infection by Pregnancy Status - United States, January 22-October 3, 2020. MMWR Morb Mortal Wkly Rep. 2020 Nov 6;69(44):1641-1647. doi: 10.15585/mmwr.mm6944e3. PMID 33151921
- [Result] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Result] Marchand G, Patil AS, Masoud AT, Ware K, King A, Ruther S, Brazil G, Calteux N, Ulibarri H, Parise J, Arroyo A, Coriell C, Cook C, Ruuska A, Nourelden AZ, Sainz K. Systematic review and meta-analysis of COVID-19 maternal and neonatal clinical features and pregnancy outcomes up to June 3, 2021. AJOG Glob Rep. 2022 Feb;2(1):100049. doi: 10.1016/j.xagr.2021.100049. Epub 2022 Jan 3. PMID 35005663
- [Result] Berthelot N, Lemieux R, Garon-Bissonnette J, Drouin-Maziade C, Martel E, Maziade M. Uptrend in distress and psychiatric symptomatology in pregnant women during the coronavirus disease 2019 pandemic. Acta Obstet Gynecol Scand. 2020 Jul;99(7):848-855. doi: 10.1111/aogs.13925. Epub 2020 Jun 3. PMID 32449178
- [Result] Davenport MH, Meyer S, Meah VL, Strynadka MC, Khurana R. Moms Are Not OK: COVID-19 and Maternal Mental Health. Front Glob Womens Health. 2020 Jun 19;1:1. doi: 10.3389/fgwh.2020.00001. eCollection 2020. PMID 34816146
- [Result] Lee CF, Hwang FM, Lin HM, Chi LK, Chien LY. The Physical Activity Patterns of Pregnant Taiwanese Women. J Nurs Res. 2016 Dec;24(4):291-299. doi: 10.1097/JNR.0000000000000158. PMID 27846101
- [Result] van Mulken MR, McAllister M, Lowe JB. The stigmatisation of pregnancy: societal influences on pregnant women's physical activity Behaviour. Cult Health Sex. 2016 Aug;18(8):921-35. doi: 10.1080/13691058.2016.1148199. Epub 2016 Mar 11. PMID 26967357
- [Result] Walasik I, Kwiatkowska K, Kosinska Kaczynska K, Szymusik I. Physical Activity Patterns among 9000 Pregnant Women in Poland: A Cross-Sectional Study. Int J Environ Res Public Health. 2020 Mar 9;17(5):1771. doi: 10.3390/ijerph17051771. PMID 32182850
- [Result] Gawrysiak MJ, Leong SH, Grassetti SN, Wai M, Shorey RC, Baime MJ. Dimensions of distress tolerance and the moderating effects on mindfulness-based stress reduction. Anxiety Stress Coping. 2016 Sep;29(5):552-60. doi: 10.1080/10615806.2015.1085513. Epub 2015 Sep 15. PMID 26293679
- [Result] Goyal M, Singh S, Sibinga EM, Gould NF, Rowland-Seymour A, Sharma R, Berger Z, Sleicher D, Maron DD, Shihab HM, Ranasinghe PD, Linn S, Saha S, Bass EB, Haythornthwaite JA. Meditation programs for psychological stress and well-being: a systematic review and meta-analysis. JAMA Intern Med. 2014 Mar;174(3):357-68. doi: 10.1001/jamainternmed.2013.13018. PMID 24395196
- [Result] Mottola MF, Davenport MH, Ruchat SM, Davies GA, Poitras VJ, Gray CE, Jaramillo Garcia A, Barrowman N, Adamo KB, Duggan M, Barakat R, Chilibeck P, Fleming K, Forte M, Korolnek J, Nagpal T, Slater LG, Stirling D, Zehr L. 2019 Canadian guideline for physical activity throughout pregnancy. Br J Sports Med. 2018 Nov;52(21):1339-1346. doi: 10.1136/bjsports-2018-100056. PMID 30337460
- [Result] Farrell T, Reagu S, Mohan S, Elmidany R, Qaddoura F, Ahmed EE, Corbett G, Lindow S, Abuyaqoub SM, Alabdulla MA. The impact of the COVID-19 pandemic on the perinatal mental health of women. J Perinat Med. 2020 Nov 26;48(9):971-976. doi: 10.1515/jpm-2020-0415. PMID 32975206
- [Result] Arzamani N, Soraya S, Hadi F, Nooraeen S, Saeidi M. The COVID-19 pandemic and mental health in pregnant women: A review article. Front Psychiatry. 2022 Sep 20;13:949239. doi: 10.3389/fpsyt.2022.949239. eCollection 2022. PMID 36203829
- [Result] Ghimire U, Papabathini SS, Kawuki J, Obore N, Musa TH. Depression during pregnancy and the risk of low birth weight, preterm birth and intrauterine growth restriction- an updated meta-analysis. Early Hum Dev. 2021 Jan;152:105243. doi: 10.1016/j.earlhumdev.2020.105243. Epub 2020 Oct 24. PMID 33190020
- [Result] Brinsley J, Schuch F, Lederman O, Girard D, Smout M, Immink MA, Stubbs B, Firth J, Davison K, Rosenbaum S. Effects of yoga on depressive symptoms in people with mental disorders: a systematic review and meta-analysis. Br J Sports Med. 2021 Sep;55(17):992-1000. doi: 10.1136/bjsports-2019-101242. Epub 2020 May 18. PMID 32423912
- [Result] Ceulemans D, Thijs I, Schreurs A, Vercammen J, Lannoo L, Deprest J, Richter J, De Catte L, Devlieger R. Screening for COVID-19 at childbirth: is it effective? Ultrasound Obstet Gynecol. 2020 Jul;56(1):113-114. doi: 10.1002/uog.22099. No abstract available. PMID 32449230
- [Result] Davis K, Goodman SH, Leiferman J, Taylor M, Dimidjian S. A randomized controlled trial of yoga for pregnant women with symptoms of depression and anxiety. Complement Ther Clin Pract. 2015 Aug;21(3):166-72. doi: 10.1016/j.ctcp.2015.06.005. Epub 2015 Jun 9. PMID 26256135
- [Result] Duchette C, Tolusso DV, Stone WJ, Blankenship MM, Tinius RA. Prenatal Yoga and Mental Health During the COVID-19 Pandemic: A Randomized-Control Trial. OBM Integr Compliment Med. 2021;6(4):10.21926/obm.icm.2104051. doi: 10.21926/obm.icm.2104051. Epub 2021 Nov 25. PMID 35287283
- See also: WHO coronavirus (COVID-19) dashboard 2020 — http://data.who.int/dashboards/covid19/cases?n=c